CLINICAL TRIAL: NCT06392789
Title: A Crossover Randomized Controlled Trial to Investigate the Acceptability and Efficacy of Cecebot, a Conversational Agent for Insomnia After Breast Cancer
Brief Title: A Conversational Agent (Cecebot) to Improve Insomnia in Stage I-III Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Hope Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RG1123931; NCI-2024-03110 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19784 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (Cecebot intervention) (Experimental): Patients receive sleep education SMS conversations and access to website content modules over 10 minutes 2-4 times per week, sleep compression SMS conversations QW, and wear activity tracker daily on weeks 1-6.
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia; Other: Internet-Based Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Text Message-Based Navigation Intervention
- GROUP II (waitlist control, Cecebot intervention) (Experimental): Patients receive sleep education SMS conversations and access to website content modules over 10 minutes 2-4 times per week, sleep compression SMS conversations QW, and wear activity tracker daily on weeks 7-12.
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia; Other: Internet-Based Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Insomnia — Receive sleep education
  Other Names: CBT-I
Other: Internet-Based Intervention — Receive access to website content modules
Other: Medical Device Usage and Evaluation — Wear activity tracker
Other: Questionnaire Administration — Ancillary studies
Other: Text Message-Based Navigation Intervention — Receive sleep compression SMS conversations
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation

SUMMARY:
This clinical trial evaluates the effect of conversational agent, Cecebot, on improving insomnia in stage I-III breast cancer survivors. Sleep disturbance ranks among the top concerns reported by breast cancer survivors and is associated with poor quality of life. Many breast cancer survivors also have decreased physical activity, which may also have a negative impact on sleep and quality of life. Cognitive behavioral therapy for insomnia (CBTi) and physical activity interventions have individually been reported to improve sleep and to have a positive impact on quality of life. Cecebot is a personalized short messaging service (SMS)-based behavioral intervention that combines CBTi and physical activity strategies that may improve sleep for breast cancer survivors.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (INTERVENTION): Patients receive sleep education SMS conversations and access to website content modules over 10 minutes 2-4 times per week, sleep compression SMS conversations once weekly (QW), and wear activity tracker daily on weeks 1-6.

GROUP II (WAITLIST CONTROL): Patients receive sleep education SMS conversations and access to website content modules over 10 minutes 2-4 times per week, sleep compression SMS conversations QW, and wear activity tracker daily on weeks 7-12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years
* Prior diagnosis of stage I-III invasive breast cancer
* Female gender
* Clinically significant insomnia symptoms, defined as a Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance 8 T-score of 55 or greater
* Insomnia complaints lasting ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, indicating ability to perform activities of daily living
* Own a smartphone with Internet connectivity
* Willing and able to complete the intervention with personal smartphone
* Proficient in speaking and reading English
* Completed breast cancer treatment within past 5 years

Exclusion Criteria:

* Prior diagnosis of restless leg syndrome, periodic leg movement disorder, narcolepsy, or rapid eye movement (REM) behavior disorder
* Current sleep apnea (treated or untreated)
* Current shiftwork
* Actively receiving chemotherapy or radiation (endocrine therapy permitted)
* Previously received CBTi therapy with a professional therapist
* Contraindications to CBTi including:

  * Active psychosis
  * Uncontrolled bipolar disorder
  * Severe depression
  * Active substance use disorder (moderate or greater severity)
* Use of prescribed sleep medication > 3 times per week
* Previously participated in user testing of the study intervention (Cecebot)
* Unwilling or unable to complete study procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment discontinuation rate | Up to week 6 of intervention
  Defined as the proportion of all treatment participants who permanently stop the intervention prior to week 6 for any reason. An all-cause discontinuation rate of 40% or less will be considered a threshold for acceptability.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to week 12
  Intervention safety will be determined by reviewing and quantifying the number of adverse events, serious events and by reviewing the type and severity of AEs attributed to study procedures among each study group.
Recruitment rates | Up to week 12
  Recruitment rate will be defined as the percentage of participants enrolled of those approached.
Enrollment rate | Up to week 12
  Enrollment rate will be defined as the percent enrolled of those eligible.
Lost to follow-up | Up to week 12
  Lost to follow-up will be defined as the percent who dropped out of those enrolled. A benchmark to determine feasibility is less than 40% loss to follow-up.
AE rate | At week 6 of intervention
  AE rate will be defined as the percentage of AEs during the intervention. The number of participants experiencing an adverse event attributable to study procedures will be compared after the first 6 weeks to identify if any detectable differences are present between the treatment group and waitlist control group.
Adherence to sleep recommendations | Up to week 12
  Adherence to sleep recommendations will be defined as the percent who reported wake time recommended by Cecebot. Participant bed times and wake times will be compared to recommendations offered by Cecebot.
Adherence to physical activity (PA) recommendation | Up to week 12
  Adherence to PA recommendations will be defined as the percent who achieved PA goals.
Data entry adherence | Up to week 12
  Data entry adherence will be defined as the percent of sleep efficiency and PA data collection forms completed.
Intervention engagement | Up to week 12
  Intervention engagement will be defined as the percent of educational modules interacted with by the user providing text-based responses.
Sleep quality and the impact of insomnia | At week 0, 6 and 12
  The Insomnia Severity Index (ISI) and daily sleep diaries will be used to assess sleep quality and the impact of insomnia. The ISI will be measured using a 5-point Likert scale of 7 questions yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Kerryn Reding, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai CS, Szewczyk W, Drerup M, Liao J, Vasbinder A, Greenlee H, Heffner JL, Yung R, Reding KW. A Personalized, Texting-Based Conversational Agent to Address Sleep Disturbance in Individuals Who Have Survived Breast Cancer: Protocol for a Pilot Waitlist Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 14;14:e62712. doi: 10.2196/62712. PMID 40658949

DOCUMENTS (1):
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT06392789/ICF_000.pdf